CLINICAL TRIAL: NCT02013271
Title: A Prospective, Multicenter, Single-Arm Trial With the Lutonix Drug Coated Balloon for Treatment of Long Lesions in Femoropopliteal Arteries
Brief Title: Lutonix® DCB for Treatment of Long Lesions in Femoropopliteal Arteries
Status: Completed | Type: Observational
Sponsor: C. R. Bard (Industry)
Responsible Party: Sponsor
Other Study IDs: CL0017-01
Record Dates: First submitted 2013-12-11; First posted 2013-12-17 (Estimated); Last update posted 2019-10-08 (Actual); Status verified 2019-10

CONDITIONS: Femoral Artery Occlusion; Femoral Arterial Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Lutonix DCB: Lutonix Paclitaxel Drug Coated Balloon
  Interventions: Device: Lutonix Paclitaxel Drug Coated Balloon (DCB)

INTERVENTIONS:
Device: Lutonix Paclitaxel Drug Coated Balloon (DCB) — Patients exposed to the DCB as part of their routine care.

SUMMARY:
To demonstrate efficacy and safety of the Lutonix® Drug Coated Balloon for treatment of long TASC II Class C and D lesions (≥ 14 cm) lesions in the SFA

DETAILED DESCRIPTION:
The study will enroll patients presenting with claudication or ischemic rest pain (Rutherford Category 2-4) and TASC II Class C or D lesions ≥14 cm in length in the native femoropopliteal artery. After successful pre-dilatation (1mm < RVD) and spot stenting (if necessary, with length minimized to mechanical defect), subjects will receive treatment with the Lutonix Drug Coated Balloon (DCB).

The primary safety and efficacy endpoint assessments are performed at 12 months. Clinical follow-up continues through a minimum of 2 years and telephone follow-up through a minimum of 3 years.

ELIGIBILITY:
Inclusion Criteria:

Clinical Criteria

1. ≥ 18 years of age;
2. Rutherford Clinical Category 2-4;
3. The subject is legally competent, has been informed of the nature, the scope and the relevance of the study, voluntarily agrees to participation and the study's provisions, is willing to provide 5-year informed consent and has duly signed the informed consent form (ICF).

   Angiographic Criteria
4. Significant (≥ 70%) stenosis or occlusion of a native femoropopliteal artery (by visual estimate) that is amenable to DCB with or without stenting;
5. TASC II Class C or D Lesions with intended target lesion treatment segment(s) cumulatively ≥14 cm in length;
6. de novo lesion(s) or non-stented restenotic lesion(s) > 90 days from prior angioplasty procedure;
7. Proximal margin of target lesion(s) starts ≥ 1 cm below the common femoral bifurcation;
8. Distal margin of target lesion(s) terminates at bifurcation of popliteal artery AND ≥1 cm above the origin of the TP trunk;
9. Target vessel diameter between ≥ 4 and ≤ 7 mm and able to be treated with available device size matrix;
10. A patent inflow artery free from significant lesion (≥ 50% stenosis) as confirmed by angiography (treatment of target lesion acceptable after successful treatment of iliac inflow artery lesions); NOTE: Successful inflow artery treatment is defined as attainment of residual diameter stenosis ≤ 30% without death or major vascular complication.
11. Successful wire crossing and pre-dilatation of the target lesion; NOTE: Use of crossing devices allowed if necessary NOTE: Bare nitinol stenting of short segments (length minimized to the mechanical defect) is required after pre-dilatation to resolve flow-limiting dissections or if deemed clinically necessary.
12. At least one patent native outflow artery to the ankle, free from significant (≥ 50%) stenosis as confirmed by angiography that has not previously been revascularized (treatment of outflow disease is NOT permitted during the index procedure);
13. No other prior vascular interventions (including contralateral limb) within 2 weeks before and/or planned 30 days after the protocol treatment.

Exclusion Criteria:

1. 1. Women who are pregnant, lactating, or planning on becoming pregnant or men intending to father children;
2. Patient is contraindicated to use Lutonix Drug Coated Balloon per the current Instructions For Use (IFU)
3. Life expectancy of < 1year;
4. Patient is currently participating in an investigational drug or other device study or previously enrolled in this study; NOTE: Enrollment in an investigational device or pharmaceutical clinical trial during the follow up period is not allowed.
5. History of stroke within 3 months;
6. History of myocardial infarction, thrombolysis or angina within 2 weeks of enrollment;
7. Prior vascular surgery of the index limb, with the exception of endarterectomy or remote common femoral patch angioplasty, separated by at least 1 cm from the target lesion;
8. Target lesion involves a previously placed stent
9. Inability to take required study medications or allergy to contrast that cannot be adequately managed with pre- and post-procedure medication;
10. No normal proximal artery segment in which duplex flow velocity can be measured;
11. Significant inflow disease. Successful treatment of inflow iliac disease allowed prior to target lesion treatment;
12. Unsuccessful crossing; NOTE: crossing devices allowed
13. Known inadequate distal outflow (> 50% stenosis of distal popliteal or all three tibial vessels), or planned future treatment of vascular disease distal to the target lesion;
14. Sudden symptom onset, acute vessel occlusion, or acute or sub-acute angiographically visible thrombus in target vessel;
15. Intended use of laser, atherectomy or cryoplasty during the index procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will enroll patients presenting with claudication or ischemic rest pain (Rutherford Category 2-4) and TASC II Class C or D lesions ≥14 cm in length in the native femoropopliteal artery. After successful pre-dilatation (1mm < RVD) and spot stenting (if necessary, with length minimized to mechanical defect), subjects will receive treatment with the Lutonix Drug Coated Balloon (DCB).
Sampling Method: Non-Probability Sample
Enrollment: 125 (Actual)
Dates: Start 2013-12 (Actual); Primary Completion 2016-05-23 (Actual); Study Completion 2018-06-13 (Actual)

PRIMARY OUTCOMES:
Overall Medical Safety | 12 Months
  Combination assessment of freedom from all-cause peri-procedural (≤30 day) death and freedom at 1 year from the following: index limb amputation (above or below the ankle) and index limb re-intervention. Success is freedom from all specified events; failure is one or more specified events occurs.
Primary Endpoint Efficacy, measured by presence of primary patency of the target lesion. Patency is assessed by a Corelab based on ultrasound images | 12 Months
  Primary Patency is defined as Freedom from Clinically-Driven Target Lesion Revascularization and from Binary Restenosis. Binary restenosis is adjudicated by the independent, blinded core laboratory based on threshold Doppler PSVR ≥ 2.5 (together with wafeform analysis & color mosaic appearance) or based on angiographic ≥ 50% diameter stenosis (if angiography is performed although not required per protocol). Clinically-Driven TLR is adjudicated by the Clincal Events Committee.

SECONDARY OUTCOMES:
Secondary Endpoint Medical Safety: Major vascular complications | ≤30 days after index procedure
  Major vascular complications will be counted:
  * Haematoma at access site >5 cm
  * False aneurysm
  * AV fistula
  * Retroperitoneal bleed
  * Peripheral ischemia/nerve injury
  * Any transfusion required will be reported as a vascular complication unless clinical indication clearly other than catheterization complication
  * Vascular surgical repair
Secondary Endpoint Medical Safety: Composite Safety | 1, 6, 12, 24, 36 months after index procedure
  Combination assessment of freedom from all-cause death and freedom from the following: index limb amputation (above or below the ankle) and index limb re-intervention. Success is freedom from all specified events; failure is one or more specified events occurs.
Secondary Endpoint Medical Safety: All-cause death | 1, 6, 12, 24, 36 months after index procedure
  Death by any cause will be counted.
Secondary Endpoint Medical Safety: Major amputation at target limb | 1, 6, 12, 24, 36 months after index procedure
  Amputations above the ankle of the target leg will be counted.
Secondary Endpoint Medical Safety: Minor amputation at target limb | 1, 6, 12, 24, 36 months after index procedure
  Amputations below the ankle of the target leg will be counted.
Secondary Endpoint Medical Safety: Target Vessel Revascularization (TVR) | 1, 6, 12, 24, 36 months after index procedure
  Repeat intervention at the target vessel will be counted.
Secondary Endpoint Medical Safety: Target Limb Reintervention | 1, 6, 12, 24, 36 months after index procedure
  Repeat intervention at the target leg will be counted.
Secondary Endpoint Efficacy: Acute Device Success | During index procedure
  Device success is defined as, a per device basis, the achievement of successful delivery and deployment of the study device(s) as intended at the intended target lesion, without balloon rupture or inflation/deflation abnormalities and a successful withdrawal of the study system. If a device is inserted into the subject but not used due to user error (e.g. inappropriate balloon length or transit time too long), this device will not be included in the device success assessment.
Secondary Endpoint Efficacy: Technical Success | During index procedure
  Technical Success of the balloon procedure is defined as successful access and deployment of the device and visual estimate of ≤ 30% diameter residual stenosis during the index procedure.
Secondary Endpoint Efficacy: Procedural Success | Until index hospitalization discharge
  Attainment of ≤ 30% residual stenosis in the treatment area by independent core lab analysis without major adverse events (defined as occurrence of death, major amputation of the target limb, target vessel or distal revascularization) during the index procedure and through the hospital stay.
Secondary Endpoint Efficacy: Primary Patency | 6, 12, 24, 36 months after index procedure
  Primary Patency is defined as Freedom from Clinically-Driven Target Lesion Revascularization and from Binary Restenosis. Binary restenosis is adjudicated by the independent, blinded core laboratory based on threshold Doppler PSVR ≥ 2.5 (together with waveform analysis & color mosaic appearance) or based on angiographic ≥ 50% diameter stenosis (if angiography is performed although not required per protocol). Clinically-Driven Target Lesion Revascularization is adjudicated by the Clinical Evenbts Committee.
Secondary Endpoint Efficacy: Secondary Patency | 6, 12, 24, 36 months after index procedure
  Secondary Patency of the target lesion is defined as the absence of binary restenosis as adjudicated by the blinded, independent core laboratory, independent of whether or not patency is re-established via an endovascular procedure.
Secondary Endpoint Efficacy: Clinically-driven Target Lesion Revascularization (TLR) | 6, 12, 24, 36 months after index procedure
  Revascularization of the target vessel with evidence of diameter stenosis >50% determined by duplex ultrasound or angiography and new distal ischemic signs (worsening ABI or worsening Rutherford Category associated with the target limb or due to clinical symptoms) OR revascularization of a target vessel with an in-lesion diameter stenosis of >70% by angiography, in the absence of the previously mentioned ischemic signs or symptoms.
Secondary Endpoint Efficacy: Target Lesion Revascularization (TLR) | 6, 12, 24, 36 months after index procedure
  A repeat revascularization procedure (percutaneous or surgical) of the original target lesion site.
Secondary Endpoint Efficacy: Change of Rutherford classification from baseline | 6, 12, 24 months after index procedure
  Patients are enrolled with a Rutherford grade of 2-4 for their target leg. The Rutherford scale is an indicator for the severity of Peripheral Vascular Disease: 0 = no symptoms, 6 = functional foot is no longer salvageable (leading to foot amputation).
Secondary Endpoint Efficacy: Change of resting Ankle Brachial Index (ABI) from baseline | 6, 12, 24 months after index procedure
  The ABI values will be recorded and compared to the baseline values. The ABI is the ratio of the blood pressure at the ankle to the blood pressure in the upper arm. A ratio of 0.9-1.3 is in the normal range. Lower ratios indicate bad blood perfusion of the leg.
Secondary Endpoint Efficacy: Change in Walking Impairment Questionnaire from baseline | 6, 12, 24 months after index procedure
  The Walking Impairment Questionnaire values will be recorded and compared to the baseline values.
  This questionnaire is a validated tool to assess walking capability in patients with Peripheral Arterial Disease in different situations. Worst possible score in this study would be 0, best possible score would be 92.
Secondary Endpoint Efficacy: Change in quality of life from baseline, as measured by EQ-5D | 6, 12, 24 months after index procedure
  The EQ-5D Questionnaire values will be recorded and compared to the baseline values.
  It is a validated questionnaire to measure the quality of life based on 5 different paremeters. Worst possible score in this study would be 0, best possible score would be 1. In addition the patient indicates her/his current health on an analog scale from 0 (worst) to 100 (best).

CONTACTS AND LOCATIONS:
Overall Officials: Martin Banyai, MD, PhD, Principal Investigator — Cantonal Hospital, Lucerne; Prof. Eric Ducasse, MD, PhD, Principal Investigator — University Hospital, Bordeaux
Locations (14):
- LKH-Univ. Klinikum Graz, Graz, Austria
- Belgium (4):
  - ZNA-Campus Middelheim, Antwerp
  - UZA Antwerp University Hospital, Edegem
  - Ziekenhuis Oost Limburg, Genk
  - AZ Groeninge, Kortrijk
- CHU Bordeaux, Talence, France
- Germany (7):
  - Ev.Krankenhaus Königin Elisabeth, Berlin
  - Asklepios Klinik St. Georg, Hamburg
  - University Clinical Center Heidelberg, Heidelberg
  - Westfälische Wilhelms-Universität Münster, Münster
  - Krankenhaus Barmherzige Brüder Regensburg, Regensburg
  - Medinos Kliniken Sonneberg, Sonneberg
  - Universitätsklinikum Tübingen, Tübingen
- Luzerner Kantonsspital, Division of Angiology, Lucerne, Switzerland

IPD SHARING:
Plan to Share IPD: No